CLINICAL TRIAL: NCT02505932
Title: Latarjet Procedure: Comparative Outcomes Study of Arthroscopic Versus Mini-open Approach With Minimum 2-year Follow-up
Acronym: Latarjet
Status: Completed | Type: Observational
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Shahnaz Klouche, MD, Physician responsible of clinical research, Hospital Ambroise Paré Paris
Other Study IDs: APR012012
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Joint Instability
Keywords: Shoulder instability
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arthroscopic Latarjet procedure: arthroscopic approach (set Depuy-Mitek, Raynham, MA)
  Interventions: Procedure: Arthroscopic Latarjet procedure
- Mini-open Latarjet procedure: mini-open approach (set Arthrex, Naples, FL)
  Interventions: Procedure: Mini-open Latarjet procedure

INTERVENTIONS:
Procedure: Arthroscopic Latarjet procedure — arthroscopic approach (set Depuy-Mitek, Raynham, MA)
  Groups: Arthroscopic Latarjet procedure
Procedure: Mini-open Latarjet procedure — mini-open approach (set Arthrex, Naples, FL)
  Groups: Mini-open Latarjet procedure

SUMMARY:
To date, use of arthroscopic procedure to perform Latarjet procedure is still technically demanding. The benefits of arthroscopic procedure need to be evaluated compared to the mini-invasive approach. The aim of this study was to assess postoperative pain during the first week, and the positioning of coracoid bone block at the anterior aspect of the glenoid. At minimum 2 years follow-up, the recurrence of shoulder instability and functional evaluation of patients according to the Western Ontario Score Index (WOSI) were assessed.

DETAILED DESCRIPTION:
This prospective comparative study was performed at two centers in 2012. Each center performed one procedure so this study was observational. All patients with a chronic anterior instability requiring bone grafting (Instability Severity Index Score>3) were included. The Latarjet procedure was performed by mini-open approach (set Arthrex, Naples, FL) in the first group, and by arthroscopic approach (set Depuy-Mitek, Raynham, MA) in the second group. The analgesic postoperative protocol was standardized (paracetamol, non-steroidal anti-inflammatory, tramadol).

ELIGIBILITY:
Inclusion Criteria:

* chronic anterior instability requiring bone grafting (Instability Severity Index Score>3)

Exclusion Criteria:

* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a chronic anterior instability requiring bone grafting (Instability Severity Index Score>3)
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Average postoperative shoulder's pain on visual analogic scale from 0 (no pain) to 10 (maximum pain) | Average during the first week

SECONDARY OUTCOMES:
Mean daily pain on visual analogic scale from 0 (no pain) to 10 (maximum pain) | Daily from day1 to day7
analgesic consumption (Number of pills) | Daily from day1 to day7
presence of postoperative discomfort symptoms (yes/no) | Daily from day1 to day7
  The presence (yes/no) of incision site pain, nausea, vomiting, vertigo, anxiety
coracoid bone block position to the anterior aspect of the glenoid on the anterior-posterior and the lateral X-ray and on CT-scan | Between 3 to 6 months follow-up
Recurrence rate of shoulder instability (number of recurrence/total number of patients) | 2-year minimal follow-up
Functional evaluation of patients | 2-year minimal follow-up
  Western Ontario Score Index (WOSI)

CONTACTS AND LOCATIONS:
Overall Officials: Shahnaz Klouche, MD, Study Director — Hospital Ambroise Paré Paris
Locations (2):
- France (2):
  - Hospital Ambroise Paré Paris, Boulogne-Billancourt
  - Clinique des Maussins, Paris